CLINICAL TRIAL: NCT06318091
Title: Nanofat Versus Platelet Poor Plasma Gel for Infraorbital Rejuvenation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS.21.09.1640
Record Dates: First submitted 2024-03-05; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Tear Trough Eyelid Deformity
Keywords: platelet poor plasma gel; nanofat; infraorbital rejuvenation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- platelet poor plasma gel group (Active Comparator): in this group, plasma gel will be injected intradermally in the dark circles.
  Interventions: Biological: platelet poor plasma gel
- nanofat group (Active Comparator): in this group, nanofat will be injected intradermally and subcutaneously in the dark circles
  Interventions: Biological: nanofat

INTERVENTIONS:
Biological: platelet poor plasma gel — injection of platelet poor plasma gel in the dark circles around the eye to rejuvenate and improve pigmentation
  Arms: platelet poor plasma gel group
Biological: nanofat — injection of nanofat in the dark circles around the eye to rejuvenate and improve pigmentation
  Arms: nanofat group

SUMMARY:
this study was conducted for evaluation of the clinical efficacy, safety, and potential side effects of platelet poor plasma gel versus nonfat injection in infraorbital rejuvenation

ELIGIBILITY:
Inclusion Criteria:

* all patients with infraorbital dark circles

Exclusion Criteria:

* pregnancy
* breast feeding
* infectious disorders

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
the degree of changes in the skin texture and homogeneity | 3 months
  the degree of changes in the skin texture and homogeneity was assessed using the five grades scale according to percentage of change in skin surface smoothness and color uniformity (1: much worse if deterioration >25%, 2: worse if deterioration <25%, 3: slightly improved if improvement <25%, 4: improved if improvement = 25%-50%, and 5: greatly improved if improvement >50%).

CONTACTS AND LOCATIONS:
Locations (1):
- Manousra University, Faculty of Medicine, Al Mansurah, Dakahlia Governorate, Egypt